CLINICAL TRIAL: NCT05138952
Title: The Mindful Media Project: Can Mindfulness Meditation Reduce for Problematic Internet Use
Brief Title: The Mindful Media Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Monash University (Other)
Collaborators: Headspace, Inc (Unknown)
Responsible Party: Principal Investigator, Rebecca Segrave, Senior Research Fellow, Monash University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 29159
Record Dates: First submitted 2021-08-10; First posted 2021-12-01 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Problematic Internet Use
MeSH Terms: interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness Meditation (Experimental): 30-day program of mindfulness meditation comprising weekly group meditation tuition and support sessions and daily app-based mediation practice.
  Interventions: Behavioral: Mindfulness Meditation

INTERVENTIONS:
Behavioral: Mindfulness Meditation — 30-day mediation program comprising:
  1. Weekly group mediation tuition and support sessions delivered online. Sessions will last 45-60 minutes and focus on mindfulness meditation theory and techniques, and trouble shooting barriers to practice and engagement.
  2. 10-minutes of daily mindfulness meditation practice with the Headspace Inc app.

SUMMARY:
Problematic Internet Use (PIU) is an emerging mental health issue. Research consistently shows that university students are disproportionately vulnerable to experiencing PIU, and that this can be linked with both poorer academic performance and mental health outcomes. Despite these adverse consequences, there has been no research to date on treatments for those experiencing PIU.

Preliminary research suggests that one promising candidate is mindfulness meditation. Mindfulness is a popular form of brain training that helps develop an ability to sit with uncomfortable thoughts and emotions, break compulsive behavioural patterns and make more mindful behavioural choices. The current proof-of-concept study aims to investigate the clinical potential of mindfulness meditation in reducing PIU severity for Australian university students who endorse moderate to severe PIU symptoms.

DETAILED DESCRIPTION:
Problematic Use of the Internet (PUI) is an umbrella term encapsulating excessive and uncontrolled engagement with internet-related activities. PIU is increasingly recognised as an emerging mental health issue. It is characterised by a perceived loss of control over internet use despite repeated attempts to regulate it, and excessive internet-specific preoccupations or urges that result in distress and life impairment. Research consistently shows that university students are disproportionately vulnerable to experiencing PIU, and that this can be linked with both poorer academic performance and mental health outcomes.

Despite these adverse consequences, there has been no research to date on treatments for those experiencing PIU. Preliminary research suggests that one promising candidate for addressing PIU is mindfulness meditation. Mindfulness is a popular form of brain training that helps develop an ability to sit with uncomfortable thoughts and emotions, break compulsive behavioural patterns and make more mindful behavioural choices.

The current study is a proof of principal investigation. The primary aim is to evaluate the efficacy of a brief mindfulness meditation intervention for PIU among Australian university students who endorse moderate to severe PIU. The study will investigate a 30 day combination of daily meditation practice using the Headspace Inc supported by weekly online group meditation tuition. In order to support participant engagement in the meditation practices, a range of behaviour change techniques will be applied. A secondary is to evaluation the efficacy of these behaviour change techniques in support engagement.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary and able to provide informed consent
* Endorse current moderate to severe PIU on IAT-10
* Currently attending an Australian university (full-time or part-time, international or domestic student)
* Ability to adhere to study procedures
* If taking psychoactive medication, have been stable on same type and dose for at least 4 weeks prior to study commencement

Exclusion Criteria:

* History of neurological illness or moderate to severe brain injury
* Severely impaired visual/auditory ability
* Diagnosed history of learning difficulty or other condition involving cognitive impairment as a primary feature.
* Lack of both verbal and written fluency in English
* Have engaged in > 10 instances of formal mindfulness meditation practice in past 12 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Change in Problematic Internet Use (PIU) severity | Change from baseline PIU severity at 1 month (post-intervention).
  10-item abbreviated Internet Addiction Test (IAT-10). Scores range from 10 to 50, with higher scores indicating increasing severity of PIU.

SECONDARY OUTCOMES:
Change in response inhibition | Baseline (0 months), Post-Intervention (1 month), Follow-Up (2-months)
  Stop Signal Task
Change in psychological distress | Change from baseline psychological distress at 1 month (post-intervention) and 2 months (one-month follow-up post intervention).
  The Depression Anxiety Stress Scale (DASS-21) consists of 21 items, 7 items per subscale: depression, anxiety and stress. For each subscale, scores can range from 0 to 42, with higher scores indicating greater severity or worse outcomes.
Change in experiential avoidance | Change from baseline experiential avoidance at 1 month (post-intervention) and 2 months (one-month follow-up post intervention).
  The Brief Experiential Avoidance Questionnaire (BEAQ) is a 15-item short form of the Multidimensional Experiential Avoidance Questionnaire. Scores can range from 15 to 90, with higher scores indicating greater experiential avoidance.
Change in trait mindfulness | Change from baseline trait mindfulness at 1 month (post-intervention) and 2 months (one-month follow-up post intervention).
  The Cognitive Affective Mindfulness Scale Revised (CAMS-R) is a 12-item scale, with scores ranging from 12 to 48. High scores indicate greater mindful qualities.
Change in psychological wellbeing | Change from baseline psychological wellbeing at 1 month (post-intervention) and 2 months (one-month follow-up post intervention).
  The Warwick-Edinburgh Mental Well-being Scale (WEMWBS) is a 14-item measure of psychological wellbeing, with scores ranging from 14 to 70. Higher scores indicate higher levels of mental wellbeing.
Change in resilience | Change from baseline resilience at 1 month (post-intervention) and 2 months (one-month follow-up post intervention).
  The Connor-Davidson Resilience Scale is a 10-item scale measuring resilience. Scores range from 0 to 40, and higher scores indicate higher resilience.
Change in social connectedness | Change from baseline social connectedness at 1 month (post-intervention) and 2 months (one-month follow-up post intervention).
  The Campaign to End Loneliness Tool is a brief 3-item measure of social connectedness. Scores range from 0 to 12, and higher scores reflect greater social connectedness.
Number of participants retained in mindfulness intervention | Post-Intervention (1 month)
  Number of participants who completed the intervention
Engagement in intervention | Post-Intervention (1 month)
  Number of meditation sessions completed

CONTACTS AND LOCATIONS:
Locations (1):
- Monash University, BrainPark, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No